CLINICAL TRIAL: NCT00858741
Title: Phase III Study of Palliative Radiotherapy for Bone Metastases Comparing Single to Multiple Fractions.
Brief Title: Palliative Radiotherapy for Bone Metastases: Single Versus Multiple Fractions.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Marilia Medicine School (Other)
Responsible Party: Gustavo Viani Arruda, Marilia Medicine School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAMEMA - BONE METASTASES
Record Dates: First submitted 2009-03-06; First posted 2009-03-10 (Estimated); Last update posted 2009-03-10 (Estimated); Status verified 2009-03

CONDITIONS: Bone Metastases; Pain
Keywords: bone metastases from any histological subtype.
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 8 Gy arm (Experimental): 8.0 Gy in 1 fraction to 8.0 Gy total dose.
  Interventions: Radiation: single fraction
- 30 Gy arm (Active Comparator): 3.0 Gy x 10 fractions to 30.0 Gy total dose in two weeks.
  Interventions: Radiation: multiple fractions

INTERVENTIONS:
Radiation: single fraction — 8 Gy x 1 fraction to 8 Gy total dose in single dose.
  Arms: 8 Gy arm
Radiation: multiple fractions — 3.0 Gy x 10 fractions to 30.0 Gy total dose in two weeks.
  Arms: 30 Gy arm

SUMMARY:
The aim of the investigators study was to determine whether 8 Gy in a single fraction provides equivalent pain and narcotic relief compared to 30 Gy in 10 fractions for patients with painful bone metastases.

The secondary objectives were to evaluate the frequency, duration of pain relief, narcotic relief, toxicity and the effect on quality of life measures for each of the two treatment arms.

DETAILED DESCRIPTION:
This prospective, phase III, randomized study was conducted by department of radiation oncology at Marilia Medicine School, São Paulo, Brazil.

Eligibility requirements included:

Age of 18 years or older, histologically proven primary malignancy of any histological type, radiographic evidence of bone metastasis, pain corresponding to the area of bone metastasis, a Karnofsky performance status of at least 40, and an estimated life expectancy of at least 1months.

Histologic diagnosis was established from needle biopsy, bone marrow biopsy, cytology, or a surgical biopsy or resection.

Radiographic evidence of bone metastasis was required and performed within 8 weeks prior to randomization. Acceptable studies included plain radiographs, radionuclide bone scans, computed tomography scans and magnetic resonance imaging. Other studies were acceptable with the approval of the principal investigator.

Eligible treatment sites were: pelvis, femur, sacrum and/or sacroiliac joints, tibia, cervical, thoracic or lumbar vertebral bodies, humerus, fibula, radius ± ulna, clavicle, sternum, scapula and púbis.

Patients had a "Worst Pain Score" of > 5 on a scale of 10 (as scored on the Brief Pain Inventory [BP]: 0 = no pain; 10 = worst possible pain) or if BPI is < 5, had be taking narcotic medications with a daily morphine equivalent dose ≥ 60 mg p.o. Patients receiving systemic therapy were eligible for this study as long as there has been no introduction of any systemic therapy within the 30 days prior to entry into this study.

The patient was ineligible if the systemic agent commences within the 30 days prior to registration. This includes hormonal therapy, chemotherapy, and immunotherapy. Patients were ineligible if the painful area had received prior radiation therapy or palliative surgery, if there was pathologic fracture or impending fracture of the treatment site, or if there was planned surgical fi xation of the bone. Patients with clinical or radiographic evidence of spinal cord or cauda equina compression and/or effacement were not eligible.

Required information before randomization included history and physical examination, Karnofsky performance status, radiographically documented bone metastases within 8 weeks before randomization, and completed Brief Pain Inventory.

RADIATION THERAPY

Treatment Plan

Arm A: 3.0 Gy x 10 fractions to 30.0 Gy total dose in two weeks. Arm B: 8.0 Gy in 1 fraction to 8.0 Gy total dose.

Simulation of treatment fields was required prior to the first treatment. Prior to the first treatment, an acceptable simulator and portal film documenting that the treatment site was adequately covered and verified by the treating radiation oncologist.

Treatment was given using megavoltage equipment with Cobalt-60 or 6-Mev photons. The minimum Source-Axis Distance (SAD) was 80 cm. All fields were treated each day. Treatment volume was including the radiographic abnormality with at least a 2 cm margin. Treatment of the entire bone is not required. Anterior and posterior parallel opposed fields were used for lumbar spine, sacrum, pelvis, and extremity sites. Equal weighting was recommended, although unequal weighting was used for the lumbar or sacral spine with a ratio of doses of 1:2 AP:PA. Dose was prescribed at mid thickness at the central axis, or at the center of target volume if unequal weighting is used. The cervical spine was treated with either parallel opposed lateral fields or with a single posterior field. When lateral fields were used, the isocenter should be at mid-thickness, with the dose prescribed to the mid-vertebral body. For a single posterior field, the dose was prescribed at a depth of 5 cm or other depth as determined from a lateral simulator film. When more than one osseous site was included into one treatment field, the treating radiation oncologist used differing field arrangements at her/his discretion, with the fields arranged to provide relatively uniform treatment of the target sites with a minimum of uninvolved normal tissues.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older, histologically proven primary malignancy of any histological type, radiographic evidence of bone metastasis, pain corresponding to the area of bone metastasis, a Karnofsky performance status of at least 40, and an estimated life expectancy of at least 1 month.
* Histologic diagnosis was established from needle biopsy, bone marrow biopsy, cytology, or a surgical biopsy or resection. Radiographic evidence of bone metastasis was required and performed within 8 weeks prior to randomization.

Exclusion Criteria:

* The patient was ineligible if the systemic agent commences within the 30 days prior to registration.
* This includes hormonal therapy, chemotherapy, and immunotherapy.
* Patients were ineligible if the painful area had received prior radiation therapy or palliative surgery, if there was pathologic fracture or impending fracture of the treatment site, or if there was planned surgical fi xation of the bone.
* Patients with clinical or radiographic evidence of spinal cord or cauda equina compression and/or effacement were not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)

PRIMARY OUTCOMES:
Pain relief

SECONDARY OUTCOMES:
duration of pain relief, narcotic relief, toxicity and the effect on quality of life measures for each of the two treatment arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Radiation Oncology Department at Marilia Medicine school, Marília, São Paulo, Brazil